CLINICAL TRIAL: NCT01163240
Title: A Cross-sectional, Multi-center, Epidemiological Study in Western and Asian Countries in Children and Adolescents With Chronic Hepatitis B
Brief Title: Epidemiological Study in Children and Adolescents With Chronic Hepatitis B
Acronym: EPIC B
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLDT600A2414
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Liver Diseases; Hepatitis, Chronic; Hepatitis, Viral, Human; Hepatitis; Virus Diseases; Digestive System Diseases; Hepatitis B, Chronic; Hepatitis B; DNA Virus Infections
Keywords: hepatitis B; HBV; chronic hepatitis B; pediatric
MeSH Terms: conditions — Liver Diseases; Hepatitis, Chronic; Hepatitis, Viral, Human; Hepatitis; Virus Diseases; Digestive System Diseases; Hepatitis B, Chronic; Hepatitis B; DNA Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- pediatric

SUMMARY:
The purpose of this study is to collect epidemiological data in children and adolescents with chronic hepatitis B(CHB), in particular data on the prevalence of HBeAg positive disease with associated ALT levels , active HBeAg negative disease and decompensated CHB in the pediatric population. Family history and history of HBV transmission is essential to assess the course of the disease and can be used to determine the best mode of treatment This information will be used to assist with the feasibility and design of studies for the Novartis clinical pediatric development program, as the current epidemiology of ediatric CHB is not accurately known in Western countries or the rest of the world making pediatric studies difficult to plan and conduct. This study forms part of the Novartis Pediatric Investigational Plan, a post marketing approval commitment to the EMEA Pediatric Committee.

ELIGIBILITY:
Inclusion criteria:

* Male or female, 2 to less than 18 years of age.
* Documented chronic hepatitis B defined by all of the following:

  * Clinical history compatible with chronic hepatitis B,Detectable serum HBsAg at the time of the study and at least one other documentation of HBsAg positive at least 6 months prior to inclusion HBeAg-positive or HBeAg-negative Serum ALT of all levels subject or subject's parent or legal guardian must be willing and able to provide written informed consent for participation in the study.

Exclusion criteria:

* Patients ≥ 18 years of age
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible patients will be identified in the treatment centers by the investigators. These patients can include those patients being referred to the practice or patients currently being seen by the investigator who are male or female, children or adolescents with chronic hepatitis B, aged 2 to < 18 years . Patients visiting the center during the 2 year enrolment period may be eligible for the study. This visit will constitute the data captured for the "current disease state" in the questionnaire. Patients will be recruited from Asian and Western countries.
Sampling Method: Probability Sample
Enrollment: 1640 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Obtain epidemiological data in children and adolescents with chronic hepatitis B that will assist the feasibility and design of studies for the Novartis telbivudine clinical pediatric development program | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (86):
- United States (5):
  - The Children's Hospital, Aurora, Colorado
  - Shands Hospital at University of Florida, Gainesville, Florida
  - Children's Hospital Boston, Boston, Massachusetts
  - Saint Vincent Healthcare Pediatric Specialty Clinics, Billings, Montana
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital de Niños Dr. Ricardo Gutierrez, Capital Federal, Buenos Aires, Argentina
- Brazil (5):
  - Hospital de Clínicas de Porto Alegre, Porto, Alegre
  - Núcleo de Estudos e Pesquisas em Hepatologia da Amazônia, Belém
  - Hospital Oswaldo Cruz - Universidade de Pernambuco, Recife
  - Instituto da Criança - HC FMUSP, São Paulo
  - Universidade de Campinas, Campinas, São Paulo
- China (17):
  - Beijing You'an Hosptial, Beijing
  - The First Affiliated Hospital of Chongqing Med. University, Chongqing
  - 1st Affliated Hospital of 3rd Military Med. Univ. of PLA, Chongqing
  - Hebei Medical University The Third Hospital, Shijiazhuang, Hebei
  - Henan Academy of Medical Pharmaceutical Sciences, Zhengzhou, Henan
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Second Xiangya Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - First Hospital University of Jilin, Changchun, Jilin
  - The First Affiliated Hospital of Medical College, Kunming, Kunming
  - The First Affiliated Hospital of Lanzhou University, Lanzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Institute of Hematol., Union Hospital, Tongji Med. College, Wuhan
  - Second Hospital of Xian Jiaotong University, Xi'an
  - Hospital of Chengdu Military Area Command, Kunming, Yunnan
- France (4):
  - Groupe Hospitalier Pellegrin - Hôpital des Enfants, Bordeaux, Aquitaine
  - Hôpital Jeanne de Flandre, Lille
  - Groupe Hospitalier Necker - Enfants Malades, Paris
  - Hôpital de Haute Pierre, Strasbourg
- Greece (5):
  - Peripheral University General Hospital of Alexandroupoli, Alexandroupoli
  - "Agia Sofia" Childrens Hospital of Athens, Athens
  - IASO Children's Hospital, Athens
  - University General Hospital of Heraklion, Heraklion, Crete
  - Childrens' General Hospital of Athens 'P&A Kyriakou', Goudi
- India (6):
  - Dr. R. K. Jain Clinic, Bhopal
  - Choithram Hospital and Research Centre, Indore
  - St. John's Medical College Hospital, Banglaore, Karna
  - Apollo Gleneagles Hospital, Kolkata
  - TNMC and BYL Nair Charitable Hospital, Mumbai
  - Maulana Azad Medical College & LNJP Hospital, New Delhi
- Italy (5):
  - Azienda Osp.-Univ. Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Istituto G. Gaslini Ospedale Pediatrico IRCCS, Genova
  - Universita degli Studi "Federico II", Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Pediatrico Bambino Gesu, Roma
- Peru (3):
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Hospital Nacional G A Yrigoyen, Lima
  - Instituto Nacional de Salud del Niño, Lima
- Philippines (4):
  - Research Institute for Tropical Medicine, City of Muntinlupa
  - Philippine General Hospital, Ermita
  - Philippine Children's Medical Center, Quezon City
  - National Kidney and Transplant Institute, Quezon City
- Poland (3):
  - Wojewodzki Spital Bydgoszcz, Bydgoszcz
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
- Romania (3):
  - "Matei Bals" Institute of Infectious Diseases, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - V. Babes Pneumology and Infectious Diseases Clin. Hosp, Craiova
- Russia (6):
  - Central Research Institute for Epidemiology of Rospotrebnadz, Moscow
  - Russian State Medical University, Moscow
  - Research Center of Children's Health, Moscow
  - Saint- Petersburg State Mtchnikov's Medical Academy, Saint Petersburg
  - Research Institute for Infectious Childhood Diseases, Saint Petersburg
  - Smolensk State Medical Academy, Smolensk
- Singapore (2):
  - National University of Singapore, Singapore
  - KK Women's and Children's Hospital, Singapore
- Spain (6):
  - Hospital Universitario San Cecilio, Granada, Andalucía
  - Hospital Sant Joan de Deu, Barcelona, Cataluña
  - Hospital Carlos III, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Hospital Universitario La Fe, Valencia
- Taiwan (4):
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veteran's General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai
- United Kingdom (5):
  - Birmingham Childrens Hospital, Birmingham
  - St James's University Hospital, Leeds
  - The Royal London Hospital, London
  - Kings College Hospital, London
  - Queen's Medical Centre, Nottingham